CLINICAL TRIAL: NCT07290283
Title: A Phase I, Randomized, Single-blind, Placebo-controlled Study to Assess the Safety, Tolerability and Pharmacokinetics of AZD3974 After Single and Multiple Ascending Dosing to Healthy Participants
Brief Title: A Study to Investigate Safety, Tolerability, and Pharmacokinetics of AZD3974 in Healthy Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: D7360C00001
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Healthy Participants
Keywords: Single ascending dose; Multiple ascending dose; Pharmacokinetics; Impact of food; First-in-human

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (28):
- Part A1 (SAD) Cohort 1: AZD3974 (Dose 1) (Experimental): Healthy participants will receive a single dose of AZD3974 - Dose 1
  Interventions: Drug: AZD3974
- Part A1 (SAD) Cohort 2: AZD3974 (Dose 2) (Experimental): Healthy participants will receive a single dose of AZD3974 - Dose 2
  Interventions: Drug: AZD3974
- Part A1 (SAD) Cohort 3: AZD3974 (Dose 3) (Food Effect Cohort) (Experimental): Healthy participants will receive two single doses of AZD3974 - Dose 3
  Interventions: Drug: AZD3974
- Part A1 (SAD) Cohort 4: AZD3974 (Dose 4) (Experimental): Healthy participants will receive a single dose of AZD3974 - Dose 4
  Interventions: Drug: AZD3974
- Part A1 (SAD) Cohort 5: AZD3974 (Dose 5) (Experimental): Healthy participants will receive a single dose of AZD3974 - Dose 5
  Interventions: Drug: AZD3974
- Part A1 (SAD) Cohort 6: AZD3974 (Dose 6) (Experimental): Healthy participants will receive a single dose of AZD3974 - Dose 6
  Interventions: Drug: AZD3974
- Part A1 (SAD) optional additional Cohort 7: AZD3974 (Experimental): Healthy participants will receive a single dose of AZD3974
  Interventions: Drug: AZD3974
- Part A1 (SAD) optional additional Cohort 8: AZD3974 (Experimental): Healthy participants will receive a single dose of AZD3974
  Interventions: Drug: AZD3974
- Part A1 (SAD) Cohort: Placebo (Placebo Comparator): Healthy participants will receive a single dose of matching placebo to AZD3974
  Interventions: Other: Placebo
- Part A1 (SAD) Cohort 3: Placebo (Food Effect Cohort) (Placebo Comparator): Healthy participants will receive two single doses of matching placebo to AZD3974
  Interventions: Other: Placebo
- Part A2 (SAD) Japanese Cohort 1: AZD3974 (Experimental): Healthy Japanese participants will receive a single dose of AZD3974
  Interventions: Drug: AZD3974
- Part A2 (SAD) Japanese Cohort 2: AZD3974 (Experimental): Healthy Japanese participants will receive a single dose of AZD3974
  Interventions: Drug: AZD3974
- Part A2 (SAD) Japanese Cohort 3: AZD3974 (Experimental): Healthy Japanese participants will receive a single dose of AZD3974
  Interventions: Drug: AZD3974
- Part A2 (SAD) optional additional Japanese Cohort 4: AZD3974 (Experimental): Healthy Japanese participants will receive a single dose of AZD3974
  Interventions: Drug: AZD3974
- Part A2 (SAD) Japanese Cohort: Placebo (Placebo Comparator): Healthy Japanese participants will receive a single dose of matching placebo to AZD3974
  Interventions: Other: Placebo
- Part A3 (SAD) Chinese Cohort 1: AZD3974 (Experimental): Healthy Chinese participants will receive a single dose of AZD3974
  Interventions: Drug: AZD3974
- Part A3 (SAD) optional additional Chinese Cohort 2: AZD3974 (Experimental): Healthy Chinese participants will receive a single dose of AZD3974
  Interventions: Drug: AZD3974
- Part A3 (SAD) Chinese Cohort: Placebo (Placebo Comparator): Healthy Chinese participants will receive a single dose of matching placebo to AZD3974
  Interventions: Other: Placebo
- Part B1 (MAD) Cohort 1: AZD3974 (Experimental): Healthy participants will receive multiple doses of AZD3974
  Interventions: Drug: AZD3974
- Part B1 (MAD) Cohort 2: AZD3974 (Experimental): Healthy participants will receive multiple doses of AZD3974
  Interventions: Drug: AZD3974
- Part B1 (MAD) Cohort 3: AZD3974 (Experimental): Healthy participants will receive multiple doses of AZD3974
  Interventions: Drug: AZD3974
- Part B1 (MAD) Cohort 4: AZD3974 (Experimental): Healthy participants will receive multiple doses of AZD3974
  Interventions: Drug: AZD3974
- Part B1 (MAD) optional additional Cohort 5: AZD3974 (Experimental): Healthy participants will receive multiple doses of AZD3974
  Interventions: Drug: AZD3974
- Part B1 (MAD) optional additional Cohort 6: AZD3974 (Experimental): Healthy participants will receive multiple doses of AZD3974
  Interventions: Drug: AZD3974
- Part Bl (MAD) Cohort: Placebo (Placebo Comparator): Healthy participants will receive multiple doses of matching placebo to AZD3974
  Interventions: Other: Placebo
- Part B2 (MAD) Japanese Cohort 1: AZD3974 (Experimental): Healthy Japanese participants will receive multiple doses of AZD397
  Interventions: Drug: AZD3974
- Part B2 (MAD) optional additional Japanese Cohort 2: AZD3974 (Experimental): Healthy Japanese participants will receive multiple doses of matching placebo to AZD3974
  Interventions: Drug: AZD3974
- Part B2 (MAD) Japanese Cohort: Placebo (Placebo Comparator): Healthy Japanese participants will receive multiple doses of matching placebo to AZD3974
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: AZD3974 — AZD3974 will be administered as an oral solution.
  Arms: Part A1 (SAD) Cohort 1: AZD3974 (Dose 1); Part A1 (SAD) Cohort 2: AZD3974 (Dose 2); Part A1 (SAD) Cohort 3: AZD3974 (Dose 3) (Food Effect Cohort); Part A1 (SAD) Cohort 4: AZD3974 (Dose 4); Part A1 (SAD) Cohort 5: AZD3974 (Dose 5); Part A1 (SAD) Cohort 6: AZD3974 (Dose 6); Part A1 (SAD) optional additional Cohort 7: AZD3974; Part A1 (SAD) optional additional Cohort 8: AZD3974; Part A2 (SAD) Japanese Cohort 1: AZD3974; Part A2 (SAD) Japanese Cohort 2: AZD3974; Part A2 (SAD) Japanese Cohort 3: AZD3974; Part A2 (SAD) optional additional Japanese Cohort 4: AZD3974; Part A3 (SAD) Chinese Cohort 1: AZD3974; Part A3 (SAD) optional additional Chinese Cohort 2: AZD3974; Part B1 (MAD) Cohort 1: AZD3974; Part B1 (MAD) Cohort 2: AZD3974; Part B1 (MAD) Cohort 3: AZD3974; Part B1 (MAD) Cohort 4: AZD3974; Part B1 (MAD) optional additional Cohort 5: AZD3974; Part B1 (MAD) optional additional Cohort 6: AZD3974; Part B2 (MAD) Japanese Cohort 1: AZD3974; Part B2 (MAD) optional additional Japanese Cohort 2: AZD3974
Other: Placebo — Placebo will be administered as an oral solution.
  Arms: Part A1 (SAD) Cohort 3: Placebo (Food Effect Cohort); Part A1 (SAD) Cohort: Placebo; Part A2 (SAD) Japanese Cohort: Placebo; Part A3 (SAD) Chinese Cohort: Placebo; Part B2 (MAD) Japanese Cohort: Placebo; Part Bl (MAD) Cohort: Placebo

SUMMARY:
The purpose of this study is to assess the safety and tolerability of AZD3974 and characterize the pharmacokinetics (PK) of AZD3974 following oral administration to healthy participants, including participants of Japanese and Chinese descent.

DETAILED DESCRIPTION:
This is a first in human, randomized, single-blind, placebo-controlled study. It consists of two parts.

Part A (single ascending dose - SAD): This study part will enroll six cohorts (plus two optional additional cohorts) of healthy participants (Part A1), three cohorts (plus one optional additional cohort) of healthy Japanese participants (Part A2) and one cohort (plus one optional additional cohort) of healthy Chinese participants (Part A3). Cohort 3 of Part A1 will be extended to evaluate the effect of food intake on the PK of AZD3974. In Part A (all cohorts), participants will receive a single dose of AZD3974 or placebo.

Part B (Multiple Ascending Dose - MAD): This study part will consist of four cohorts (plus two optional additional cohorts) of healthy participants (Part B1) and one cohort (plus one optional additional cohort) of healthy Japanese participants (Part B2). In all Part B cohorts, participants will receive multiple doses of AZD3974 or placebo.

Both Part A and Part B will comprise of:

* A Screening Period of maximum 28 days
* A Dosing session during which participants will receive the study intervention at study specific time points.
* Follow-up Period of 7 days post last-dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female (of non-childbearing potential) participants with suitable veins for cannulation or repeated venipuncture at the Screening Visit.
* All females must have a negative pregnancy test. Females of non-childbearing potential must be confirmed via post-menopausal status or documentation of irreversible surgical sterilization at the Screening Visit.
* Sexually active fertile male participants with partners of childbearing potential must adhere to the contraception methods.
* Have a body mass index between 18 and 32 kg/m2 inclusive and weigh at least 50 kg at Screening.
* For healthy Japanese cohorts (Part A2 and Part B2): healthy male and female participants are to be Japanese (eg, natives of Japan or Japan Americans), defined as having both parents and 4 grandparents who are Japanese. This includes second and third generation participants of Japanese descent whose parents or grandparents are living in a country other than Japan.
* For healthy Chinese cohort (Part A3): healthy male and female Chinese participants for whom both parents and 4 grandparents are Chinese. This includes second and third generation participants of Chinese descent whose parents or grandparents are living in a country other than China.

Exclusion Criteria:

* History of any clinically important disease or disorder which, may either put the participant at risk because of participation in the study, or influence the results or the participant's ability to participate in the study.
* History or presence of gastrointestinal, hepatic, or renal disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Any clinically important illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of study intervention.
* Any abnormal laboratory values, vital signs, or any clinically important abnormalities in clinical chemistry, hematology, or urinalysis results.
* Any positive result on Screening for serum hepatitis B and C viruses and human immunodeficiency virus.
* Any clinically important abnormalities in rhythm, conduction, or morphology of the resting 12 lead electrocardiography at Screening and/or admission to the Clinical Unit .
* Known or suspected history of alcohol or drug abuse or excessive intake of alcohol.
* Positive screen for drugs of abuse, or alcohol, or cotinine.
* History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity.
* Participants who have previously received AZD3974.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 176 (Estimated)
Dates: Start 2025-12-10 (Actual); Primary Completion 2026-10-14 (Estimated); Study Completion 2026-10-14 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) and serious adverse events (SAEs) | Part A: Upto Day 7; Part A1 Cohort 3: Upto Day 10; Part B: Upto Day 14
  To assess the safety and tolerability of AZD3974 following oral administration of single and multiple ascending doses in healthy participants, including Chinese and Japanese participants

SECONDARY OUTCOMES:
Part A and Part B: Plasma concentrations of AZD3974 | Part A: Day 1 to Day 2; Part B: Day 1 to Day 9
  To characterize the plasma concentrations of AZD3974 following single and multiple ascending doses in healthy participants, including Chinese and Japanese participants.
Part A1-Cohort 3: Plasma concentrations of AZD3974 | Day 1 to Day 4
  To assess the impact of food (fed) on the single-dose plasma concentrations of AZD3974
Part A and Part B: Urine concentrations of AZD3974 | Part A: Day 1; Part B: Day 1 and Day 7
  To characterize the urine concentration of AZD3974 following single and multiple ascending doses in healthy participants, including Chinese and Japanese participants.
Part A1-Cohort 3: Urine concentrations of AZD3974 | Day 1 and Day 3
  To assess the impact of food (fed) on the single-dose urine concentrations of AZD3974
Part A and Part B: Area under concentration-curve from time 0 to the last quantifiable concentration (AUClast) | Part A: Day 1 to Day 2; Part B: Day 1 to Day 9
  To characterize the PK of AZD3974 following single and multiple ascending doses in healthy participants, including Chinese and Japanese participants
Part A1-Cohort 3: Area under concentration-curve from time 0 to the last quantifiable concentration (AUClast) | Day 1 to Day 4
  To assess the impact of food (fed) on the single-dose PK of AZD3974
Part A: Area under concentration-time curve from time 0 to infinity (AUCinf) | Day 1 to Day 2
  To characterize the PK of AZD3974 following single ascending doses in healthy participants, including Chinese and Japanese participants
Part A1-Cohort 3: Area under concentration-time curve from time 0 to infinity (AUCinf) | Day 1 to Day 4
  To assess the impact of food (fed) on the single-dose PK of AZD3974
Part A and Part B: Maximum observed drug concentration (Cmax) | Part A: Day 1 to Day 2; Part B: Day 1 to Day 9
  To characterize the PK of AZD3974 following single and multiple ascending doses in healthy participants, including Chinese and Japanese participants
Part A1-Cohort 3: Maximum observed drug concentration (Cmax) | Day 1 to Day 4
  To assess the impact of food (fed) on the single-dose PK of AZD3974
Part A and Part B: Time to reach maximum observed concentration (tmax) | Part A: Day 1 to Day 2; Part B: Day 1 to Day 9
  To characterize the PK of AZD3974 following single and multiple ascending doses in healthy participants, including Chinese and Japanese participants
Part A1-Cohort 3: Time to reach maximum observed concentration (tmax) | Day 1 to Day 4
  To assess the impact of food (fed) on the single-dose PK of AZD3974
Part A and Part B: Terminal elimination half-life (t½λz) | Part A: Day 1 to Day 2; Part B: Day 1 to Day 9
  To characterize the PK of AZD3974 following single and multiple ascending doses in healthy participants, including Chinese and Japanese participants
Part A1-Cohort 3: Terminal elimination half-life (t½λz) | Day 1 to Day 4
  To assess the impact of food (fed) on the single-dose PK of AZD3974
Part A and Part B: Apparent total body clearance (CL/F) | Part A: Day 1 to Day 2; Part B: Day 1 to Day 9
  To characterize the PK of AZD3974 following single and multiple ascending doses in healthy participants, including Chinese and Japanese participants
Part A1-Cohort 3: Apparent total body clearance (CL/F) | Day 1 to Day 4
  To assess the impact of food (fed) on the single-dose PK of AZD3974
Part A and Part B: Apparent volume of distribution based on the terminal phase (Vz/F) | Part A: Day 1 to Day 2; Part B: Day 1 to Day 9
  To characterize the PK of AZD3974 following single and multiple ascending doses in healthy participants, including Chinese and Japanese participants
Part A1-Cohort 3: Apparent volume of distribution based on the terminal phase (Vz/F) | Day 1 to Day 4
  To assess the impact of food (fed) on the single-dose PK of AZD3974
Part A and Part B: Individual and cumulative amount of unchanged drug excreted into urine from time t0 to time tlast [Ae(0-last)] | Part A: Day 1; Part B: Day 1 and Day 7
  To characterize the PK of AZD3974 following single and multiple ascending doses in healthy participants, including Chinese and Japanese participants
Part A1-Cohort 3: Individual and cumulative amount of unchanged drug excreted into urine from time t0 to time tlast [Ae(0-last)] | Day 1 and Day 3
  To assess the impact of food (fed) on the single-dose PK of AZD3974
Part A and Part B: Individual and cumulative percentage of dose excreted unchanged in urine from time t0 to tlast [fe(0-last)] | Part A: Day 1; Part B: Day 1 and Day 7
  To characterize the PK of AZD3974 following single and multiple ascending doses in healthy participants, including Chinese and Japanese participants
Part A1-Cohort 3: Individual and cumulative percentage of dose excreted unchanged in urine from time t0 to tlast [fe(0-last)] | Day 1 and Day 3
  To assess the impact of food (fed) on the single-dose PK of AZD3974
Part A and Part B: Renal clearance (CLR) | Part A: Day 1; Part B: Day 1 and Day 7
  To characterize the PK of AZD3974 following single and multiple ascending doses in healthy participants, including Chinese and Japanese participants
Part A1-Cohort 3: Renal clearance (CLR) | Day 1 and Day 3
  To assess the impact of food (fed) on the single-dose PK of AZD3974
Part A and Part B: Mean Residence Time (MRT) | Part A: Day 1 to Day 2; Part B: Day 1 to Day 9
  To characterize the PK of AZD3974 following single and multiple ascending doses in healthy participants, including Chinese and Japanese participants.
Part A1-Cohort 3: Mean Residence Time (MRT) | Day 1 to Day 4
  To assess the impact of food (fed) on the single-dose PK of AZD3974
Part A and Part B: Time delay between drug administration and the first observed concentration (tlag) | Part A: Day 1 to Day 2; Part B: Day 1 to Day 9
  To characterize the PK of AZD3974 following single and multiple ascending doses in healthy participants, including Chinese and Japanese participants.
Part A1-Cohort 3: Time delay between drug administration and the first observed concentration (tlag) | Day 1 to Day 4
  To assess the impact of food (fed) on the single-dose PK of AZD3974
Part A and Part B: Time of last quantifiable concentration (tlast) | Part A: Day 1 to Day 2; Part B: Day 1 to Day 9
  To characterize the PK of AZD3974 following single and multiple ascending doses in healthy participants, including Chinese and Japanese participants.
Part A1-Cohort 3: Time of last quantifiable concentration (tlast) | Day 1 to Day 4
  To assess the impact of food (fed) on the single-dose PK of AZD3974
Part A and Part B: Individual and cumulative amount of unchanged drug excreted into urine from time t1 to time t2 [Ae(t1 t2)] | Part A: Day 1; Part B: Day 1 and Day 7
  To characterize the PK of AZD3974 following single and multiple ascending doses in healthy participants, including Chinese and Japanese participants.
Part A1-Cohort 3: Individual and cumulative amount of unchanged drug excreted into urine from time t1 to time t2 [Ae(t1 t2)] | Day 1 and Day 3
  To assess the impact of food (fed) on the single-dose PK of AZD3974
Part A and Part B: Individual and cumulative percentage of dose excreted unchanged in urine from time t1 to time t2 - [fe(t1-t2)] | Part A: Day 1; Part B: Day 1 and Day 7
  To characterize the PK of AZD3974 following single and multiple ascending doses in healthy participants, including Chinese and Japanese participants.
Part A1-Cohort 3: Individual and cumulative percentage of dose excreted unchanged in urine from time t1 to time t2 - [fe(t1-t2)] | Day 1 and Day 3
  To assess the impact of food (fed) on the single-dose PK of AZD3974
Part A and Part B: Cumulative amount of unchanged drug excreted into urine (Aeinf) | Part A: Day 1; Part B : Day 1 and Day 7
  To characterize the PK of AZD3974 following single and multiple ascending doses in healthy participants, including Chinese and Japanese participants.
Part A1-Cohort 3: Cumulative amount of unchanged drug excreted into urine (Aeinf) | Day 1 and Day 3
  To assess the impact of food (fed) on the single-dose PK of AZD3974
Part B: Area under concentration time curve in the dosing interval (AUCtau) | Day 1 to Day 9
  To characterize the PK of AZD3974 following multiple ascending doses in healthy participants, including Japanese participants
Part B: Observed lowest concentration before the next dose is administered: (Ctrough) | Day 1 to Day 9
  To characterize the PK of AZD3974 following multiple ascending doses in healthy participants, including Japanese participants.
Part B: Accumulation ratio for AUC calculated as steady State AUCτ/First Dose AUCτ (Rac AUC) | Day 1 to Day 9
  To characterize the PK of AZD3974 following multiple ascending doses in healthy participants, including Japanese participants
Part B: Accumulation ratio for Cmax calculated as steady State Cmax/First Dose Cmax (Rac Cmax) | Day 1 to Day 9
  To characterize the PK of AZD3974 following multiple ascending doses in healthy participants, including Japanese participants.
Part B: Temporal change parameter calculated as steady State AUCτ/First Dose AUCinf (TCP) | Day 1 to Day 9
  To characterize the PK of AZD3974 following multiple ascending doses in healthy participants, including Japanese participants.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Research Site, Glendale, California
  - Research Site, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/